CLINICAL TRIAL: NCT00582088
Title: A Phase 2 Open-Label, Safety and Immunogenicity Study of Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI-GSD 205 When Used as a Booster After TC-83 Primary Immunization in Healthy Adults At-Risk for Exposure to Virulent Venezuelan Equine Encephalomyelitis Virus
Brief Title: Safety and Immunogenicity of Venezuelan Equine Encephalomyelitis Vaccine (VEE C-84) as a Booster to VEE TC-83
Acronym: VEE C-84
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-14350; FY06-27 (Other: SIP)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Venezuelan Equine Encephalomyelitis
Keywords: Encephalitis, Viral Infections, Neurologic diseases, Alphavirus Infections, VEE
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine; Encephalitis; Virus Diseases; Nervous System Diseases; Alphavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): VEE C-84 - Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI-GSD 205
  Interventions: Biological: VEE C-84

INTERVENTIONS:
Biological: VEE C-84 — Subjects will receive a 0.5 mL subcutaneous injection in the upper outer aspect of arm; maximum of four boosters in 1 year if titer <1:20.

SUMMARY:
The study is designed to assess the safety and immunogenicity of Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI GSD 205, as a booster vaccination.

DETAILED DESCRIPTION:
Study Objectives:

Primary:

To assess safety of Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI GSD 205, as a booster vaccination as a single dose or a three-dose series, and To assess immunogenicity of Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI GSD 205, as a booster vaccination as a single dose or a three-dose series

Secondary:

To assess incidence of VEE infection in C-84 boosted personnel.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* VEE PRNT80 < 1:20 before immunization.
* (females) Negative urine pregnancy test on the same day before vaccination. Not planning pregnancy for 3 months.
* Actively enrolled in the SIP.
* At risk for exposure to virulent VEE virus (with up-to-date risk assessment).
* Previous TC-83 vaccination
* Up-to-date (within 1 year) physical examination/tests.
* Sign and date the approved informed consent.
* Willing to return for all follow-up visits.
* Agree to report adverse event (AE) up to 28 days after vaccination.

Exclusion Criteria:

* Over age of 65 years
* Clinically significant abnormal lab results including evidence of Hepatitis C, Hepatitis B carrier state, or elevated liver function tests.
* History of immunodeficiency or current treatment with immunosuppressive medication.
* (females) Currently breastfeeding.
* Confirmed human immunodeficiency virus (HIV) titer.
* Any known allergies to components of the vaccine.
* A medical condition that in the judgment of the Principal Investigator (PI) would impact subject safety (i.e-vaccination and or exposure to another alphavirus).
* Administration of any vaccine within 28 days of C-84.
* Any unresolved AEs resulting from a previous immunization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (ITT) | Day 28 after each booster dose
  Frequency of the following adverse events will be evaluated for all intent-to-treat subjects: headache, myalgia, fever, fatigue, sore throat, erythema, tenderness, and warmth.
Immunogenicity: TC-83 with PRNT80 ≥ 1:20 | Between Days 28 and 35 after each booster dose
  Number of initial responders to TC-83 with PRNT80 ≥ 1:20 after C-84 booster dose.
Immunogenicity: TC-83 with PRNT80 ≥ 1:20 | 12-15 months after booster dose
  Number of initial responders to TC-83 with PRNT80 ≥ 1:20 after C-84 booster dose.
Immunogenicity: TC-83 with PRNT80 < 1:20 | Between Days 28 and 35 after each booster dose
  Number of initial responders to TC-83 who are non-responders (PRNT80 < 1:20) to C-84 booster dose.
Immunogenicity: TC-83 with PRNT80 < 1:20 | 12-15 months after vaccination
  Number of initial responders to TC-83 who are non-responders (PRNT80 < 1:20) to C-84 booster dose.
Immunogenicity: TC-83 with PRNT80 ≥ 1:20 after three booster doses | After three booster doses
Immunogenicity: TC-83 with PRNT80 ≥ 1:20 12- 15 months after first booster dose | 12- 15 months after first booster dose
Immunogenicity: PRNT80 ≥ 1:20 after 1 dose | After 1 dose
  Number of rollovers from past C-84 booster study with PRNT80
  ≥ 1:20 after 1 dose.
Immunogenicity: PRNT80 ≥ 1:20 12-15 months post dose for new C-84 Protocol. | 12-15 months post dose for new C-84 Protocol

SECONDARY OUTCOMES:
VEE disease among vaccinated subjects who achieved a PRNT80 ≥ 1:20. | Length of the study
  The number of confirmed cases of VEE disease among vaccinated subjects who achieved a PRNT80
  ≥ 1:20.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Cardile, DO, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States